CLINICAL TRIAL: NCT03565861
Title: A Phase 1, Randomized , Double Blind, Single Ascending Dose Study to Investigate Safety, Tolerability and PK of NP10679 in Healthy Adults
Brief Title: Safety and Pharmacokinetics of NP10679 in Normal Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurop Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: NP10679-001
Record Dates: First submitted 2018-05-29; First posted 2018-06-21 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Safety Issues

STUDY DESIGN:
Intervention Model Description: Adaptive design of placebo and up to six escalating doses of NP10679
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Placebo (Placebo Comparator): Placebo intravenous 30 minute infusion on day 1
  Interventions: Drug: Placebo
- NP10679 5 mg (Experimental): NP10679 5 mg intravenous infusion on day 1
  Interventions: Drug: NP10679
- NP10679 15 mg (Experimental): NP10679 15 mg intravenous infusion on day 1
  Interventions: Drug: NP10679
- NP10679 50 mg (Experimental): NP10679 50 mg intravenous infusion on day 1
  Interventions: Drug: NP10679
- NP10679 100 mg (Experimental): NP10679 100 mg intravenous infusion on day 1
  Interventions: Drug: NP10679
- NP10679 200 mg (Experimental): NP10679 200 mg intravenous infusion on day 1
  Interventions: Drug: NP10679
- NP10679 300 mg (Experimental): NP10679 300 mg intravenous infusion on day 1
  Interventions: Drug: NP10679

INTERVENTIONS:
Drug: Placebo — Intravenous vehicle
  Arms: Placebo
Drug: NP10679 — NP10679
  Arms: NP10679 100 mg; NP10679 15 mg; NP10679 200 mg; NP10679 300 mg; NP10679 5 mg; NP10679 50 mg

SUMMARY:
This study assesses the safety, tolerability and pharmacokinetics of NP10679 when delivered intravenously in escalating dose levels in comparison to placebo.

DETAILED DESCRIPTION:
NP10679 is a pH dependent inhibitor of the GluN2B subtype of the NMDA receptor. Compounds of this drug class are hypothesized to be beneficial in a number of central nervous system disorders, including brain ischemia associated with subarachnoid hemorrhage, severe pain, major depression and substance abuse disorders. This study uses a double blind, adaptive design approach to evaluate the safety, tolerability and pharmacokinetics of a single dose of NP10679 when delivered intravenously in up to six escalating dose levels in comparison to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18 to 55 years
* Ability to understand the requirements of the study, provide written informed consent, abide by the study restrictions, and agree to return for the required assessments.
* If of child bearing potential (both men and women) must agree to use 2 forms of contraceptive methods for the duration of study.

Exclusion Criteria:

* Clinical laboratory values greater than or equal to 2 times the upper limit of normal.
* Recent history (within 2 yrs) or current tobacco use.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2018-09-02 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events as a measure of safety and tolerability | 8 days
  Observed side effects and alteration in laboratory values.

SECONDARY OUTCOMES:
Plasma concentration of parent drug | 4 days
  Cmax after administration.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Zaczek, Ph.D., Study Chair — Neurop Inc.; Paolo DePetrillo, Principal Investigator — Pharmaron CPC
Locations (1):
- Pharmaron CPC, Baltimore, Maryland, United States